CLINICAL TRIAL: NCT06684691
Title: The Effect of an Escape Room Simulation on Post-mortem Care Training for Nursing Students: a Randomised Controlled Trial
Brief Title: The Effect of an Escape Room Simulation on Post-mortem Care Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Gül ŞAHİN KARADUMAN, Asst. Prof., Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Date: 10.09.2924 No:2024-436
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Simulation Training; Game-Based Learning; Nursing Care
Keywords: Escape room; Simulation; Nursing student; Education; Post-mortem care
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel group trial
Masking Description: There is no blinding because of the nature of the simulation method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): The escape room game will be applied to the students in the group 1 after the theoretical training.
  Interventions: Other: Intervention group
- Group 2 (Other): The escape room game will not be applied to the students in the group 2 after the theoretical training.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — The escape room game will be applied to the students in the intervention group after the theoretical training.
  Arms: Group 1
Other: Control group — The escape room game will not be applied to the students in the control group after the theoretical training.
  Arms: Group 2

SUMMARY:
Simulated escape room games create an active learning environment to increase students' motivation and participation and encourage learning while developing skills. Therefore, this study examines the effectiveness of simulated escape room games in nursing students' post-mortem care education.

DETAILED DESCRIPTION:
To meet the emotional and physical needs of the individual living in the last days of life, the nurse must have the necessary knowledge, skills, and understanding. For this reason, post-mortem care has an important place in the nursing education curriculum. To increase student motivation and include them in the learning process in clinical skills laboratory environments, game strategies have been frequently used in education in recent years. The "escape room" game has emerged as a new pedagogical method to provide interactive teaching. The use of interactive teaching and games in health education has a positive effect on the learning process.

ELIGIBILITY:
Inclusion Criteria:

* Being 4th grade nursing student

Exclusion Criteria:

* Not willing to participate the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
Knowledge | 5 week
  Postmortem Care Knowledge Test
Self-Efficacy | 5 week
  End of Life and Post-Death Self-Efficacy Scale for Nursing Students

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Gulhane Faculty of Nursing, Ankara, Please Select One, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
At the end of the study, we can share the study.

REFERENCES:
- [Derived] Basak T, Demirtas A, Sahin Karaduman G, Duman S, Cerit B. The Effect of an Escape Room Simulation on Postmortem Care Training For Nursing Students: A Randomized Controlled Trial. J Hosp Palliat Nurs. 2026 Jan 1;28(1):E17-E23. doi: 10.1097/NJH.0000000000001166. Epub 2025 Sep 17. PMID 41373097